CLINICAL TRIAL: NCT00375908
Title: Umbilical Cord Blood Proteomic Analysis and Neonatal Brain Injury
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Ernest M. Graham, M.D., Associate Professor, Johns Hopkins University
Other Study IDs: 861
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Hypoxia-Ischemia, Brain; Periventricular Leukomalacia
Keywords: Neonatal Encephalopathy; Hypoxic-Ischemic Brain Injury; Umbilical Cord Blood; Proteomics
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Leukomalacia, Periventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to compare the proteomic analysis of umbilical venous blood from neonates with brain injury to gestational age matched noninjured controls. After delivery an umbilical arterial gas and a 10 ml umbilical venous sample are obtained, then the remainder of the cord blood is discarded. The investigators plan to use this cord blood that would otherwise be discarded to perform our proteomic analysis. The investigators will use up to 20 ml of cord blood per delivery. This will be a 5 year study during which time the investigators hope to analyze 450 infants at Johns Hopkins Hospital and Bayview Medical Center. The investigators will obtain an umbilical venous sample from infants born at < 34 weeks gestation. For infants born at > 34 weeks the investigators will obtain an umbilical venous sample for any infant suspected to be at risk for neurologic injury by having a diagnosis of chorioamnionitis during labor, nonreassuring fetal heart rate tracing at the time of delivery, or a 5 minute Apgar < 7. For the infants born at < 34 weeks the brain injured infants will be compared to gestational age matched controls without brain injury. For the infants born at > 34 weeks, each infant later confirmed to have neurologic morbidity will be compared to a gestational age matched noninjured control. The investigators hope to use proteomic analysis to determine if there are measurable differences in protein expression between the 2 groups.

DETAILED DESCRIPTION:
We will draw up to 20 ml of umbilical venous blood at the time of delivery from infants born at < 34 weeks gestation, and for any infant born at > 34 weeks suspected to be at risk for neurologic morbidity by having intrapartum chorioamnionitis, nonreassuring fetal heart tracing prior to delivery, or a 5 minute Apgar < 7. For each infant born at > 34 weeks later confirmed to have neurologic morbidity by head ultrasound or EEG we will draw cord blood from a gestational age matched control without intrapartum infection or nonreassuring fetal heart tracing prior to delivery. At the time of delivery an umbilical arterial gas and umbilical venous sample for a type and screen, RPR and hematocrit are routinely drawn. The remainder of the cord blood is discarded. After the routinely done arterial blood gas and umbilical venous blood sample are obtained the remainder of the umbilical cord blood, which would otherwise be discarded, will be collected using a 23 gauge or larger needle into a heparinized tube. The sample will be centrifuged for 10 minutes and the plasma layer separated. The sample will be placed into 1.5 ml eppendorf tubes in 500 ul aliquots. Proteomic techniques including mass spectrometry, 2-dimensional electrophoresis, and chromatography, will be used to analyze the proteome from the brain injured and control groups. Specific proteins will be identified, and differences in expression compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Less than 34 weeks gestational age or more than 34 weeks with a risk factor for brain injury such as chorioamnionitis, nonreassuring fetal heart rate tracing, metabolic acidosis, or hypotonia at birth.

Exclusion Criteria:

* Major congenital or chromosomal abnormalities in fetus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study looked at umbilical cord blood from normal neonates and neonates with risk factors for neurological injury.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Umbilical Cord Blood Proteomic Analysis and Neonatal Brain Injury | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ernest M Graham, M.D., Principal Investigator — Johns Hopkins Medicine, Dept Gyn-Ob
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States